CLINICAL TRIAL: NCT00133224
Title: A Phase III Randomized, Open-Label Study of Docetaxel in Combination With CG1940 and CG8711 Versus Docetaxel and Prednisone in Taxane-Naïve Patients With Metastatic Hormone-Refractory Prostate Cancer With Pain
Brief Title: Docetaxel in Combination With GVAX ® Immunotherapy Versus Docetaxel and Prednisone in Prostate Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual and treatment with CG1940/CG8711 stopped due to IDMC recommendation.
Sponsor: Cell Genesys (Industry)
Responsible Party: Cell Genesys, Inc., Cell Genesys, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-0034; VITAL-2
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Prostate Cancer
Keywords: Advanced Prostate Cancer; HRPC; Prostate; Cancer; Metastatic; Hormone-refractory; GVAX; Chemotherapy; Taxotere; Docetaxel; Prednisone; Vaccine; Allogeneic cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Drug Therapy; Docetaxel; Prednisone

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine
- 2 (Other)
  Interventions: Drug: Chemotherapy (docetaxel and prednisone)

INTERVENTIONS:
Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine — Immunotherapy allogeneic GM-CSF secreting cellular vaccine
  Arms: 1
Drug: Chemotherapy (docetaxel and prednisone) — Chemotherapy (docetaxel and prednisone)
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the duration of survival between patients receiving docetaxel in combination with the GVAX® vaccine for prostate cancer versus patients receiving docetaxel and prednisone treatment in patients with prostate cancer who no longer respond to hormone therapy, who have documented metastases with pain. Patients may have had up to one prior non-taxane chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of or clinical history consistent with adenocarcinoma of the prostate
* Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy
* Detectable metastases
* ECOG performance status ≤2 (Performance status of 3 if due to bone pain)
* Any Gleason score
* Only one prior treatment with systemic chemotherapy
* No prior treatment with gene therapy
* No prior immunotherapy for prostate cancer
* Taxane naïve
* Experiencing cancer-related pain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Survival | 0

SECONDARY OUTCOMES:
Time to disease progression. Time to pain progression. | 0

CONTACTS AND LOCATIONS:
Locations (115):
- United States (43):
  - Alaska Clinical Research Center, Anchorage, Alaska
  - St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Loma Linda University, Loma Linda, California
  - Onocology Care Medical Associates, Los Angeles, California
  - Desert Hematology Oncology Medical Group, Rancho Mirage, California
  - San Bernardino Urology Associates, San Bernardino, California
  - Kaiser Permanente Medical Group Dept. of Oncology Research, San Diego, California
  - Sharp Healthcare, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF Mt. Zion Cancer Center, San Francisco, California
  - Cancer Research & Prevention Center, Soquel, California
  - Cancer Center and Department of Medicine, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Jupiter Hematology & Oncology Associates, Jupiter, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Peachtree Hematology & Oncology Consultants, PC, Atlanta, Georgia
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Medical & Surgical Specialists, Galesburg, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - General Clinical Research Center University of Michigan, Ann Arbor, Michigan
  - Billings Clinic, Billings, Montana
  - Hematology & Oncology Consultants P.C., Omaha, Nebraska
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Oncology, Albuquerque, New Mexico
  - North Shore Hematology Oncology Associates P.C., East Setauket, New York
  - NYU Clinical Cancer Center, New York, New York
  - Presbyterian Hospital Center for Cancer Research, Charlotte, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Oncology/Hematology, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Center for Oncology Research & Treatment, PA, Dallas, Texas
  - Dallas Oncology Consultants, Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - Mobley Research Center, Houston, Texas
  - Northwest Cancer Center, Houston, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Seattle Cancer Care Alliance, Univ. of Washington, Seattle, Washington
- Belgium (6):
  - Ziekenhuis Netwerk Antwerpen - AZ Middelheim, Antwerp
  - V.Z.W. Imelda Ziekenhuis, Bonheiden
  - AZ Groeninge, Kortrijk
  - CHU de Liège - Hôpital du Sart Tilman, Liège
  - Heilig-Hartziekenhuis Campus Wilgenstraat, Roeselare
  - Regionaal Ziekenhuis Sint Trudo, Sint-Truiden
- Canada (2):
  - Centre Hospitalier de L'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier Universite de Sherbrooke, Sherbrooke, Quebec
- France (15):
  - Centre Regional de lutte contre le cancer Paul Papin, Angers
  - Centre Francois Baclesse, Caen
  - Institut Jean Godinot, Oncologie Medicale, Cedex
  - Centre Jean Perrin Centre Régional de lutte contre le cancer d'Auvergne, Clermont-Ferrand
  - Centre Rene Gauducheau - Site Hospitalier Nord, Nantes
  - Centre Antoine Lacassagne - Centre Regional de lutte contre le cancer, Nice
  - CHU Saint Louis, Paris
  - Hopital Saint Joseph Site Saint Michel, Paris
  - Hopital Cochin, Paris
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Rene Dubos, Pontoise
  - Clinique Armoricaine de Radiology, Saint-Brieuc
  - Hopital Civil, Strasbourg
  - CHU Bretonneau, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (8):
  - Universitatsklinikum Aachen, Aachen
  - Charite Campus Mitte, Berlin
  - Krankenhaus Am Urban, Berlin
  - Universitatsklinikum Carl Gustav Carus An Der, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt am Main
  - Urologische Klinik und Poliklinik der Johannes Gutenberg Universitat Mainz, Mainz
  - Klinikum Mannheim, Mannheim
  - Urologische Klinik und Poliklinik, München
- Italy (11):
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Azienda Ospedaliera Maggiore della Carita, Novarra
  - Azienda Ospedaliera di Parma, Parma
  - Azienda Ospedaliero Universitaria (A.O.U.) Pisana-Ospedale S. Chiara, Pisa
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Presidio Ospedaliero di Sassari-Ospedale SS. Anunziata, Sassari
  - A.S.O. San Giovanni Battista di Torino, Turin
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Academisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Poland (11):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Bialystok
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Bytom
  - Katedra i Klinika Onkologii i Radioterapli, Gdansk
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Katowice
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie Oddzial w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 1 Przemienienia Panskiego AM w Poznaniu, Poznan
  - Wojewodzki Szpital Specjalistyczny w Siedlcach, Siedlce
  - Wojewodzki Szpital Specjalistyczny Oddzial Urologii, Słupsk
  - Szpital Kliniczny Dzieciatka Jezus - Centrum Leczenia Obrazen, Warsaw
  - Centrum Onkologii Instytut im. Marii Sklodowskiej- Curie, Warsaw
- Sweden (3):
  - Universitetssjukhuset i Lund, Lund
  - University Hospital MAS (UMAS), Malmo
  - Akademiska Sjukhuset i Uppsala, Uppsala
- United Kingdom (13):
  - Addenbrookes Hospital, Cambridge
  - Royal Surrey County Hospital, Guildford
  - St. James University Hospital, Leeds
  - Lincoln County Hospital, Lincoln
  - Royal Marsden Hospital, London
  - Department of Oncology Hammersmith Hospital, London
  - Christie Hospital Manchester, Manchester
  - Clatterbridge Centre For Oncology, Metropolitan Borough of Wirral
  - Mount Vernon Hospital, Middlesex
  - Nottingham City Hospital, Nottingham
  - Rosemere Cancer Centre, Royal Preston Hospital, Preston
  - Scunthorpe General Hospital, Dept of Oncology, Scunthorpe
  - Royal Marsden Academic Urology Unit, Sutton

REFERENCES:
- [Derived] Michael BD, Syndikus I, Clark A, Baborie A. Diffuse primary leptomeningeal melanocytosis in a patient receiving a novel cancer cell vaccine for prostate cancer. BMJ Case Rep. 2010 May 4;2010:bcr11.2009.2495. doi: 10.1136/bcr.11.2009.2495. PMID 22736604